CLINICAL TRIAL: NCT06282003
Title: Protective Lung Ventilation Procedure During General Anesthesia Reduces the Incidence of Pulmonary Complications After Abdominal Surgery, Possibly
Brief Title: Protective Anesthesiological Management Procedure Imposes Control on Respiratory Comlications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masa Kontic (Other Government)
Collaborators: Prof.Dinko Tonković, MD, PhD Head of Department of Anesthesiology, Reanimatology and Intensive Care Medicine and Pain Therapy, University Hospital Centre Zagreb (Unknown); Assist. Prof. Slavica Sović, MD, PhD Department of Medical Statistics, Epidemiology and Medical Informatics, School of Public Health Andrija Štampar (Unknown); Prof. Goran Šimić, MD, PhD Professor of Neuroscience and Anatomy, Chair, Department of Neuroscience, Croatian Institute for Brain Research, University of Zagreb (Unknown); Prof. Anamarija Jazbec, Faculty of Forestry and Wood Technology, University of Zagreb (Unknown); Marijan Jedvaj, MD Anesthesiologist and ICU physician (Consultant), Head of Department of Anesthesia and IC, General Hospital Zabok (Unknown)
Responsible Party: Sponsor-Investigator, Masa Kontic, Croatian Health Insurance Fund, Croatian Health Insurance Fund
Organization: Croatian Health Insurance Fund (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 380-59-10106-21-111/148
Record Dates: First submitted 2024-01-30; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Well-Being, Psychological
Keywords: general anaesthesia; intraoperative complications; postoperative complications; lung recruitment procedure therapeutic positive-pressure ventilation
MeSH Terms: conditions — Psychological Well-Being; Intraoperative Complications; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: A crossover design should be utilized in addition to the randomization procedure to properly address outcome variability. This study was a prospective, single-center, randomized controlled, patient- and evaluator-blinded clinical investigation with a two-arm parallel design to assess the advantage of the protective (optimized) ventilation procedure (PV group of patients) compared to the conventional (standard) method of lung ventilation (CV) during general anesthesia.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional ventilation procedure (Active Comparator)
  Interventions: Procedure: The procedure of protective lung ventilation
- The protective lung ventilation procedure (Experimental): In the PV group, laung protective ventilation also included the procedure of opening the alveoli (recruitment maneuver, RM). RM was performed twice. The first instance occurred following the administration of anesthesia, with a FiO2 value of 50% (0.5). The second instance took place shortly before extubation. RM consisted of maintaining an airway pressure of 40-45 kPa for 40 s, which keeps the collapsed alveoli open and corresponds to maximum spontaneous inhalation. The specified pressure of PEEP during RM refers to conditions where hemodynamic stability. PEEP was set at 7 kPa, but just before the extubation and awakening, patients were switched to spontaneous breathing the PEEP was set to 10 kPa. There was no additive effect of positive pressure, just an addition of 3 kPa positive airway pressure was applied to keep current alveoli open continuously and possibly recruit some new ones in that short period, which corresponds to the stochastic model of respiration.
  Interventions: Procedure: The procedure of protective lung ventilation

INTERVENTIONS:
Procedure: The procedure of protective lung ventilation — The procedure of protective lung ventilation in the PV group of patients included preoxygenation with 60% oxygen in a mixture with air for 3 min, which maintained the target peripheral oxygen saturation at values above 94%, endotracheal intubation, volume-controlled mechanical ventilation, a tidal volume of 6 ml per kg of body weight. Normocarbia during the protective ventilation procedure was maintained by adjusting the minute ventilation, which is the product of the respiratory rate (12-14 breaths per minute) and the tidal volume set to 6 ml/kg of body weight. The most critical variable for the adjustment was the inhalation-exhalation ratio of 1:2, which ensured adequate oxygenation and removal of carbon dioxide during anesthesia. Identically as in the PV group, the target peripheral saturation was kept above 94% with an inspiratory oxygen concentration of 50% and peak airway pressure values of up to 40 kPa.

SUMMARY:
Anesthetic effects, surgery, and invasive mechanical intubation can impair respiratory function during general anesthesia. The risk factors for postoperative pulmonary complications (PPCs) include the type of surgery and duration, ventilation-perfusion discrepancy, and the presence of pain. Mitigating PPCs under anesthesia is a goal, but effective strategies are yet to be defined. Conventional ventilation (CV) procedure uses more inspired oxygen during pre-oxygenation and anesthesia maintenance. The protective lung ventilation (PV) procedure, on the other hand, includes high positive end-expiratory pressure, lung recruitment maneuver, oxygen saturation levels above 94%, lower inspired oxygen levels, and continuous positive airway pressure before the tube is removed. In this study, 56 consecutive patients undergoing abdominal surgery were randomly assigned, with 30 in the CV and 23 in the PV group, while 3 were lost during the follow-up. We concluded that the implementation of protective lung ventilation strategies has the potential to reduce the occurrence of PPCs, recommending these strategies be adopted as the standard practice in general anesthesia.

DETAILED DESCRIPTION:
Additionally, despite accumulated knowledge and careful monitoring, sometimes an anesthesiologist is still unable to entirely avoid the occurrence of atelectasis, a common phenomenon observed during general anesthesia. Altogether, it can be concluded that the effects of mechanical ventilation and oxygenation over an extended period are not yet well understood, particularly regarding the impact of reducing tidal volume and using higher PEEPs. This study was a prospective, single-center, randomized controlled, patient- and evaluator-blinded clinical investigation with a two-arm parallel design to assess the advantage of the protective (optimized) ventilation procedure (PV group of patients) compared to the conventional (standard) method of lung ventilation (CV) during general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* the inclusion criteria were as follows:
* subject status according to the American Society of Anesthesiologists Association classification
* ASA 1 (normal healthy patients, i.e. patients without associated comorbidities) or ASA 2 (patients with mild systemic disease, such as well-controlled hypertension), normal heart and lung function, both sexes,
* non-smokers, normal X-ray findings for heart and lungs,
* age 18-65 years,
* planned operation of medial laparotomy for colorectal cancer with a minimum duration of anesthesia of at least one hour,
* signed informed consent.
* In the case of hypertension in ASA 2 patients enrolled in the study, by examining the self-monitoring diary for the past three months (as described in Gropper et al., 2019), there was no increase in systolic pressure more than 20 mmHg from the average daily value and no increase in diastolic arterial pressure more than 10 mmHg from the average daily value.
* In the case of diabetes type II in ASA 2 patients enrolled in the study, the HbA1c values were not higher than 7% while taking oral hypoglycemic drugs and having a regulated diet. The patients enrolled also had no complications or episodes of hypoglycemia in the past three months, as described by Gropper et al., 2019.
* In the case of thyroid disease in ASA 2 patients enrolled in the study, values of TSH, fT3, and fT4 in the period up to 6 months since the last examination were normal.

Exclusion Criteria:

* ASA 4 status
* terminal renal illness
* cardiac status NYHA III i NYHA IV
* at home oxygenotherapy during 16 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Oxygentation | 10 months
  The primary outcome was the incidence of early preoperative pulmonary complications (within the first 5 postoperative days).

CONTACTS AND LOCATIONS:
Locations (1):
- General hospital Zabok, Zabok, Croatia

IPD SHARING:
Plan to Share IPD: Undecided